CLINICAL TRIAL: NCT01549340
Title: Evaluation of Patient Initiation and Persistence With Advised Allergen Immunotherapy
Brief Title: Retrospective Record Review of Adults and Children Advised for Allergen Immunotherapy (MK-7243-022)
Status: Completed | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 7243-022
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Perennial Allergic Rhinitis; Seasonal Allergic Rhinitis
Keywords: Rhinitis; Allergen immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Rhinitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Allergic Rhinitis (AR): Patients in a private allergy practice who were diagnosed with AR, with or without asthma, and advised to consider AIT between January 2005 and June 2011 and whose medical records were retrospectively reviewed.

SUMMARY:
The purpose of this study is to determine the proportion of participants that initiate allergen immunotherapy (AIT) upon the recommendation of their physician and the proportion of participants that persist with their AIT throughout the recommended course.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AR with or without allergic conjunctivitis (AC)
* Documented provider-to-patient or parent discussion of AIT as a treatment option

Exclusion Criteria:

* Participants receiving AIT as an AR treatment without documented provider-to-patient or parent discussion of AIT as a treatment option
* Participants receiving immunotherapy for insect sensitivities only
* AIT started before 2005

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were managed by physicians in a large allergy practice, recommended for AIT between 2005 and 2011 and identified by their electronic health records.
Sampling Method: Non-Probability Sample
Enrollment: 8790 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

REFERENCES:
- [Derived] Anolik R, Schwartz AM, Sajjan S, Allen-Ramey F. Patient initiation and persistence with allergen immunotherapy. Ann Allergy Asthma Immunol. 2014 Jul;113(1):101-7. doi: 10.1016/j.anai.2014.04.008. Epub 2014 May 9. PMID 24814759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study involved a retrospective record review of patients in a private allergy and asthma practice who were recommended to receive allergen immunotherapy (AIT) to treat their allergic rhinitis (AR) by their physician between January 2005 and June 2011.
Groups:
- Participants With AR: Participants with AR whose records were retrospectively reviewed
Period: Overall Study
Arm/Group | Participants With AR
Started | 8790 (Advised to receive AIT)
Started AIT | 3182
Completed | 385 (Completed 5 years of AIT)
Not Completed | 8405

BASELINE CHARACTERISTICS:
Arm/Group | Participants With AR
Number analyzed (Participants) | 8790
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (16.1)
Gender [Count of Participants; unit: Participants]
  Female | 4439
  Male | 4351

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Advised to Start AIT Who Elected Subcutaneous Immunotherapy (SCIT) Shots or Sublingual Immunotherapy (SLIT) Drops
Description: The percentage of participants who were advised by their physician to start AIT and elected to initiate AIT was calculated. AIT initiation was broken down by type of AIT initiated (SCIT or SLIT).
Time Frame: Up to 5 years
Population: The analysis population consisted of those participants with AR who were advised by their physician to receive AIT to treat their AR.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With AR
Number analyzed (Participants) | 8790
percentage of participants
  Elected SCIT | 28.2
  Elected SLIT | 8.0

2. Primary Outcome: Percentage of Participants Who Initiated SCIT or SLIT and Completed 5 Years of Treatment
Description: The percentage of participants who initiated SCIT or SLIT and completed 5 years of treatment was calculated. Duration of SCIT or SLIT was based on dates when allergy extract prescriptions were refilled. If extract refills continued past the recommended time for therapy (e.g. 5 years from the start of therapy), the participant was deemed successful in completing the recommended course. If the extract refills stopped prior to the end of the recommended time for therapy, but the last refill occurred within 6 months of the recommended time for therapy, this participant was deemed successful in completing the recommended course.
Time Frame: At 5 years
Population: The analysis population consisted of those participants with AR who were advised by their physician to receive AIT to treat their AR and who initiated AIT.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With AR
Number analyzed (Participants) | 3182
percentage of participants
  Completed 5 years of SCIT (n=2481) | 10.8
  Completed 5 years of SLIT (n=701) | 2.6

3. Primary Outcome: Duration of Treatment With SCIT or SLIT
Description: The mean duration in years of SCIT or SLIT treatment for all participants with AR who initiated SCIT or SLIT was calculated. Duration of SCIT or SLIT was based on dates when allergy extract prescriptions were refilled.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Participants With AR
Number analyzed (Participants) | 3182
years
  SCIT | 2.4 (1.8)
  SLIT | 1.9 (1.4)

4. Primary Outcome: Reason for Discontinuation of SCIT or SLIT More Than 6 Months Before Completion of the Recommended Course
Description: The reason for discontinuation of SCIT or SLIT treatment more than 6 months before completion of the recommended course of therapy was recorded. The percentage of participants whose records were reveiwed and who discontinued SCIT or SLIT due to different reasons was calculated.
Time Frame: Up to 5 years
Population: The analysis population consisted of those participants with AR who were advised by their physician to receive AIT to treat their AR, who initiated and subsequently discontinued AIT, and had their charts reviewed for the reason for discontinuation.
Measure: Number; unit: percentage of participants
Groups:
- Participants With AR Who Discontinued SCIT: Participants with AR whose records were retrospectively reviewed and discontinued SCIT
- Participants With AR Who Discontinued SLIT: Participants with AR whose records were retrospectively reviewed and discontinued SLIT
Arm/Group | Participants With AR Who Discontinued SCIT | Participants With AR Who Discontinued SLIT
Number analyzed (Participants) | 785 | 231
percentage of participants
  No reason documented | 67 | 69
  Adverse event | 7 | 4
  Lack of efficacy | 1 | 3
  Financial | 4 | 4
  Other reason | 21 | 20

5. Secondary Outcome: Percentage of Participants With a Co-morbidity of Asthma Who Initiated SCIT or SLIT
Description: The percentage of participants who had AR and asthma and initiated SCIT or SLIT was calculated.
Time Frame: Up to 5 years
Population: The analysis population consisted of those participants with AR and asthma who were advised by their physician to receive AIT to treat their AR and who initiated SCIT or SLIT.
Measure: Number; unit: percentage of participants
Groups:
- Participants With AR and Asthma: Participants with AR and asthma whose records were retrospectively reviewed
Arm/Group | Participants With AR and Asthma
Number analyzed (Participants) | 3175
percentage of participants
  Initiated SCIT | 25.2
  Initiated SLIT | 8.7

6. Secondary Outcome: Duration of SCIT or SLIT Treatment for Participants With AR and Asthma or AR Alone
Description: The mean duration in years of SCIT or SLIT treatment for all participants with AR and asthma and for all participants with AR only was calculated. Duration of SCIT or SLIT treatment was based on dates when allergy extract prescriptions were refilled.
Time Frame: Up to 5 years
Population: The analysis population consisted of those participants with AR and asthma or AR alone who were advised by their physician to receive AIT to treat their AR and who initiated AIT.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Participants With AR and Asthma: Participants with AR and asthma who elected AIT and whose records were retrospectively reviewed
- Participants With AR Alone: Participants with AR alone who elected AIT and whose records were retrospectively reviewed
Arm/Group | Participants With AR and Asthma | Participants With AR Alone
Number analyzed (Participants) | 1076 | 2106
years
  SCIT | 2.4 (1.77) | 2.4 (1.82)
  SLIT | 2.1 (1.50) | 1.8 (1.37)

ADVERSE EVENTS:
Description: Adverse events leading to discontinuation were reviewed in this retrospective chart review, but clinical and laboratory adverse events were not collected prospectively.
Arm/Group | Participants With AR
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall be notified and have a right to timely and prior review of public disclosures of the results, including without limitation, disclosures at research seminars, lectures and professional meetings and submission of papers for publication.